CLINICAL TRIAL: NCT00005429
Title: Clinical Cardiovascular Outcomes of African-Americans
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4347; R03HL051001 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To examine clinical cardiovascular outcomes of African Americans.

DETAILED DESCRIPTION:
BACKGROUND:

It has been well recognized for years that the survival rates among African-Americans with chronic diseases are reduced compared to their white counterparts. Recently attention has focussed on racial disparities in survival with chronic cardiovascular diseases. Prior to the widespread availability of coronary arteriography, African-Americans were thought to have a very low incidence of coronary artery disease. These findings appear to be inconsistent with the now generally accepted view that the coronary artery disease mortality rate is nearly equal in United States Black and white men and is increased in Black women as compared to white women.

Howard University and Howard University Hospital provided a unique environment for studying the clinical cardiovascular outcomes of African-Americans, in light of its history. That is, due to the influx of blacks into the District of Columbia in 1862, Freedmen's Hospital (which is now known as Howard University Hospital) was established for their care. Howard University Hospital has had an admissions profile with greater than 95 percent African-Americans for the past century

DESIGN NARRATIVE:

The study used previously collected data to: 1) examine the trends in mortality rates at Howard University Hospital, based on discharge status, between 1986 - 1992, for selected cardiovascular diseases; 2) compare cardiovascular mortality rate trends between Howard University Hospital and the National Hospital Discharge data; 3) examine cardiovascular co- morbidity experiences using a severity of illness index at Howard University Hospital compared to National data by race/ethnicity, geographic location and hospital bed size; and 4) identify a cohort of cardiovascular patients retrospectively based on repeated discharge data at Howard University Hospital, to analyze survival data.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1996-03 (Actual)